CLINICAL TRIAL: NCT00797368
Title: Manual Therapy and Exercise Versus Home Exercises in the Management of Patients Status Post Ankle Sprain: A Multi-Center Randomized Clinical Trial
Brief Title: Manual Therapy and Exercise Versus Home Exercises in the Management of Patients Status Post Ankle Sprain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Franklin Pierce University (Other)
Responsible Party: Principal Investigator, Joshua Cleland, DPT, OCS, Professor, Franklin Pierce University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIC0828
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Ankle Sprain
Keywords: ankle sprain; manual therapy; exercise; physical therapy; Patients who have sustained an inversion ankle sprain
MeSH Terms: conditions — Ankle Injuries; Motor Activity | interventions — Musculoskeletal Manipulations; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual Therapy and Exercise (Experimental): Manual Therapy and Exercise
  Interventions: Other: Manual Therapy and Exercise
- Home Exercise (Active Comparator): Home Exercise
  Interventions: Other: Home exercises

INTERVENTIONS:
Other: Manual Therapy and Exercise — Manual Therapy and Exercise
  Arms: Manual Therapy and Exercise
Other: Home exercises — Home exercises
  Arms: Home Exercise

SUMMARY:
A recent study has demonstrated that a physical therapist directed exercise program did not result in greater reductions in disability and pain when compared to a home exercise program. However, no manual therapy procedures were incorporated into the physical therapy treatment program despite recent evidence suggesting that thrust and non-thrust manual therapy techniques may be beneficial in reducing disability, pain and improving gait. Therefore, the purpose of this study is to compare the effectiveness of a physical therapy management approach consisting of manual therapy and exercise to a home program of exercise only. The investigators hypothesize that the group receiving manual therapy and exercise will have better outcomes.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

* A combination of physical examination and self-report measures will be used to assess the patient's potential eligibility according to each inclusion/exclusion criterion.
* The following inclusion criteria will be used to determine eligibility for this study:

  * Primary complaint of ankle pain, status post inversion ankle sprain.
  * The investigators decided to include patients with both acute and chronic ankle sprains since our previous work has shown that patients from both stage have exhibited positive benefits with manual therapy.66
  * Age between 16-60 years old
  * NPRS score > 3 points (average score) over past 24 hrs.
  * Does not meet criteria for needing radiographs per the Ottawa Ankle Rules
* The following exclusion criteria will be used to determine ineligibility for this study:

  * Red flags noted in the patient's Medical Screening Questionnaire (i.e. tumor, fracture, RA, osteoporosis, prolonged history of steroid use, severe vascular disease, etc.)
  * Prior surgery to the distal tibia, fibula, ankle joint, or rearfoot region (proximal to the base of the metatarsals).
  * Grade III ankle sprain (as defined by the West Point Ankle Sprain Grading System and/or tenderness along the anterior medial malleolus as described by,51 fracture, or other absolute contraindications to manual therapy.
  * Insufficient English language skills to complete all questionnaires
  * Inability to comply with treatment and follow-up schedule

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2008-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Foot and Ankle Ability Measure | 4-weeks and 6-months

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | 4-weeks and 6-months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Colorado University, Denver, Colorado
  - Regis University, Denver, Colorado
  - Concord Hospital, Concord, New Hampshire

REFERENCES:
- [Derived] Cleland JA, Mintken PE, McDevitt A, Bieniek ML, Carpenter KJ, Kulp K, Whitman JM. Manual physical therapy and exercise versus supervised home exercise in the management of patients with inversion ankle sprain: a multicenter randomized clinical trial. J Orthop Sports Phys Ther. 2013;43(7):443-55. doi: 10.2519/jospt.2013.4792. Epub 2013 Apr 29. PMID 23628755